CLINICAL TRIAL: NCT02162888
Title: A Phase I, Bioequivalence Study to Evaluate Two Formulations of Bendamustine (BDM) Hydrochloride (HCl) Administered to Cancer Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eagle Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: EGL-BDM-C-1301
Record Dates: First submitted 2014-06-04; First posted 2014-06-13 (Estimated); Last update posted 2021-06-07 (Actual); Status verified 2021-06

CONDITIONS: Cancer Which Has Either Progressed or Relapsed After Standard Therapy, or for Which no Curative or Standard Therapy is Appropriate
MeSH Terms: interventions — Bendamustine Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Eagle-BDM; Teva-BDM; Teva-BDM (Other): Eagle-BDM: IV Teva-BDM: IV
  Interventions: Drug: Test Product (Bendamustine)
- Teva-BDM; Eagle-BDM;Teva-BDM (Other): Eagle-BDM: IV Teva-BDM: IV
  Interventions: Drug: Test Product (Bendamustine)
- Teva-BDM, Teva-BDM, Eagle-BDM (Other): Eagle-BDM: IV Teva-BDM: IV
  Interventions: Drug: Test Product (Bendamustine)

INTERVENTIONS:
Drug: Test Product (Bendamustine)

SUMMARY:
The purpose of this study is to demonstrate that a new formulation of an Bendamustine (BDM) Hydrochloride (HCl) is bioequivalent (BE) (similar) to the commercially available product in patients with cancer.

DETAILED DESCRIPTION:
This is an open-label, randomized, crossover, Phase I study intended to demonstrate the BE, and safety and tolerability profile of 2 formulations of BDM HCl administered to cancer patients: Eagle-BDM and Teva-BDM Histologically confirmed diagnosis of any malignant disease (solid tumors and hematologic malignancies are eligible) for which no curative or standard therapy is appropriate.

At the end of the study, patients may be enrolled into an open-label extension (OLE) study (Study EGL-BDM-C-1301-OLE), at the discretion of the investigator.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of any malignant disease for which no curative or standard therapy is appropriate.
* Bone Marrow Function and Blood Chemistry results within protocol limits

Exclusion Criteria:

* CLL
* HIV
* Presence of brain metastases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2013-11; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
To demonstrate bioequivalent area under the time concentration curve (AUC) for both drug products | Participants will be in the study for up to 65 days
  Each patient will receive 3, single doses of study medication in a 56 day treatment period (2 cycles of 28 days each). Medication will be administered on Cycle 1, Day 1; Cycle 1, Day 2; and Cycle 2, Day 1. Each patient will receive 1 dose of Eagle-BDM and 2 doses of Teva-BDM in 3 randomly assigned, varying treatment sequences(Eagle-BDM, Teva-BDM, Teva-BDM; Teva-BDM, Eagle-BDM, Teva-BDM; or Teva-BDM, Teva-BDM, Eagle-BDM). Pharmacokinetic assessments will be performed.

CONTACTS AND LOCATIONS:
Locations (10):
- United States (10):
  - Oncology Institute of Hope and Innovation, Long Beach, California
  - Cancer Center of Kansas, Wichita, Kansas
  - Regional Cancer Care Associates, Cherry Hill, New Jersey
  - Penn State University Hershey Medical Center, Hershey, Pennsylvania
  - Greenville Hospital System University Medical Center, Greenville, South Carolina
  - Texas Oncology, Fort Worth, Texas
  - Scott & White Healthcare, Temple, Texas
  - Virginia Oncology Associates, Norfolk, Virginia
  - Evergreen Hematology & Oncology, Spokane, Washington
  - Yakima Valley Memorial Hospital/North Star Lodge, Yakima, Washington

REFERENCES:
- [Result] Cheung EM, Edenfield WJ, Mattar B, Anthony SP, Mutch PJ, Chanas B, Smith M, Hepner A. Safety and Pharmacokinetics of Bendamustine Rapid-Infusion Formulation. J Clin Pharmacol. 2017 Nov;57(11):1400-1408. doi: 10.1002/jcph.942. Epub 2017 May 31. PMID 28561902